CLINICAL TRIAL: NCT06792578
Title: Association Between Surgical Start Time and Postoperative Mortality, Morbidity, and Healthcare Utilization in Elective Non-cardiac Surgeries: a Retrospective, Single-center Study Using Propensity Score Matching
Brief Title: Surgical Start Time and Prognosis
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji-Hoon Sim, Assistant Professor, Asan Medical Center
Other Study IDs: AMC 2022-0755
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2022-06

CONDITIONS: Surgery; Non Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Procedure: Surgical Start Time — This intervention focuses on the retrospective analysis of the association between surgical start times (morning, afternoon, and nighttime) and postoperative outcomes in non-cardiac surgeries. The study evaluates how the timing of surgery impacts mortality, complications, transfusion rates, and ICU admissions in a tertiary hospital setting

SUMMARY:
Surgical start times significantly impacted mortality, morbidity, and resource utilization, particularly in high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients who underwent non-cardiac surgery

Exclusion Criteria:

* Emergency surgeries
* Cadaver surgeries
* Transplantation surgeries
* Patients with incomplete or missing data, such as follow-up information, operation start times, or laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients aged 18 years or older who underwent elective non-cardiac surgeries at a tertiary hospital. Patients with emergency surgeries, incomplete data on surgical start times, or missing follow-up information were excluded from the analysis. The study focuses on evaluating the impact of surgical start times (morning, afternoon, and nighttime) on postoperative outcomes, including mortality, complications, and ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 291051 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
30-Day Postoperative Mortality | 30 days post-surgery
  "The primary outcome measure is the incidence of 30-day postoperative mortality in patients undergoing non-cardiac surgeries. Mortality is defined as death occurring within 30 days following the surgery. The study aims to evaluate the association between surgical start times (morning, afternoon, and nighttime) and the risk of mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The dataset used and/or analyzed during the current study is available from the corresponding author upon reasonable request.